CLINICAL TRIAL: NCT03508219
Title: POLish Bifurcation Optimal Treatment Strategy Study for Left Main Bifurcation Percutaneous Coronary Intervention (PCI)
Acronym: POLBOS-LM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19; safety concerns; funding
Sponsor: ECRI bv (Industry)
Collaborators: Cardialysis BV (Industry); Balton Sp.zo.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRI-010
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Coronary Stenosis
Keywords: Coronary Artery Disease (CAD); Percutaneous Coronary Intervention (PCI); Left Main Bifurcation
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BiOSS LIM C (Experimental): The treatment strategy consists of contemporary PCI of the left-main bifurcation, using the BiOSS LIM C stent system, following diagnostic angiography demonstrating significant distal unprotected left main disease and local Heart Team discussion applying the anatomic SYNTAX Score.
  Interventions: Device: BiOSS LIM C

INTERVENTIONS:
Device: BiOSS LIM C — The BiOSS LIM C (Bifurcation Optimization Stent System, Balton, Warsaw, Poland). The BiOSS LIM C is a dedicated bifurcation stent covered with a mixture of a biodegradable polymer and the antiproliferative substance sirolimus. BiOSS LIM C will be used for treatment of the Left-Main bifurcation, according to its instructions for use.
  The Alex-Plus cobaltchromium sirolimus eluting stent (Balton, Warsaw, Poland) will be used for treatment of distal left-main side branches according to its instructions for use (i.e. proximal segments of the left anterior descending and left circumflex arteries as well as the ramus intermedius if the latter vessel is part of a trifurcation).
  All other lesions (other than left-main bifurcations) will be treated with XIENCE family everolimus-eluting coronary stent systems.
  Other Names: ALEX Plus; XIENCE

SUMMARY:
The primary objective of this study is to study the safety and efficacy of the BiOSS LIM C with respect to Patient oriented Composite Endpoint (PoCE) at 12 months in a "real world" left-main bifurcation population and as compared with a prespecified performance goal.

ELIGIBILITY:
Inclusion Criteria:

* Patient has distal unprotected Left-Main coronary artery (ULMCA) disease with angiographic diameter stenosis (DS) ≥50% requiring revascularization.
* Left-Main Medina classification 100, 110, 101, 011, 010, 111
* Clinical and anatomic eligibility for PCI as agreed by the local Heart Team including anatomic SYNTAX Score (<33).
* Distal left main reference vessel diameter ≥3.0 mm and ≤5.5 mm. All target lesions must be located in a native coronary artery.
* Patient with silent ischemia, chronic stable angina or stabilized acute coronary syndromes with normal cardiac biomarker values
* Able to understand and provide informed consent and comply with all study procedures including follow-up

Exclusion Criteria:

* Prior PCI of the left main bifurcation at any time prior to enrollment
* Currently participating in another trial and not yet at its primary endpoint.
* Prior PCI of any other (non left main bifurcation) coronary artery lesion within 6 months (<6 months) prior to enrollment.
* Left-Main Medina classification 001.
* Any segment of the left main bifurcation (distal left main, ostial Left Anterior Descending Artery (LAD) or ostial Left Circumflex Artery (LCX) presenting with a chronic total occlusion, or containing a visible thrombus.
* Excessive angulation of the left main bifurcation (i.e. an angulation >90° between proximal LAD and proximal LCX)
* Direct stenting of the left main bifurcation
* Prior Coronary Artery Bypass Surgery (CABG) at any time prior to enrollment
* Patient requiring or may require additional surgery (cardiac or non-cardiac) within one year
* Ongoing myocardial infarction or recent myocardial infarction with cardiac biomarker levels still elevated.
* Known renal insufficiency (e.g. serum creatinine >2.5mg/dL, or creatinine clearance ≤30mL/min, or patient on dialysis).
* Known contraindication or hypersensitivity to sirolimus, everolimus, cobalt-chromium, or to medications such as aspirin, heparin, bivalirudin, and all of the following four medications: clopidogrel bisulfate, ticlopidine, prasugrel, ticagrelor.
* Patients unable to tolerate, obtain or comply with dual antiplatelet therapy for at least 12 months.
* Patient is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential).
* Concurrent medical condition with a life expectancy of less than 12 months.
* The patient is unwilling/not able to return for outpatient clinic at 12 month follow-up.
* Currently participating in another trial and not yet at its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gil, Prof., Principal Investigator — Central Clinical Hospital of the Ministry of Interior in Warsaw
Locations (15):
- France (4):
  - Research Centre FRA-001, Aix-en-Provence
  - Research Centre FRA-004, Bron
  - Research Centre FRA-003, Grenoble
  - Research Centre FRA-002, Saint-Denis
- Italy (3):
  - Research Centre ITA-001, Naples
  - Research Centre ITA-002, Ragusa
  - Research Centre ITA-003, Syracuse
- Poland (8):
  - Research Centre PL-006, Katowice
  - Research Centre PL-007, Krakow
  - Research Centre PL-004, Olsztyn
  - Research Centre PL-005, Poznan
  - Research Centre PL-001, Warsaw
  - Research Centre PL-008, Warsaw
  - Research Centre PL-002, Zabrze
  - Research Centre PL-003, Zabrze

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Rationale and design of the POLBOS LM study — https://eurointervention.pcronline.com/article/treatment-with-a-dedicated-bifurcation-sirolimus-eluting-cobalt-chromium-stent-for-distal-left-main-coronary-artery-disease-rationale-and-design-of-the-polbos-lm-study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol aimed for 260 patients; 130 were enrolled in 14 interventional cardiology centers in Europe: Poland (8), Italy (2), and France (4). The last patient enrolled signed the informed consent on April 15th 2020, and underwent the index procedure on April 16th 2020. The last 12-month follow-up visit took place on 15 April 2021.
Period: Overall Study
Arm/Group | BiOSS LIM C
Started | 130
Completed | 121
Not Completed | 9
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 4
Not completed — Missed visit | 2

BASELINE CHARACTERISTICS:
Population: The intended sample size was 260, but the study was terminated prematurely and only 130 participants were enrolled.
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age reported in years after birth
  Years | 67.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex reported as binary, male and female
  Participants
    Female | 27
    Male | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 130
  Unknown or Not Reported | 0
Syntax Score [Mean (Standard Deviation); unit: Scores on a scale] — The SYNTAX (Synergy between Percutaneous Coronary Intervention with TAXUS and Cardiac Surgery) Score measures the anatomical complexity of coronary artery disease based on angiographic findings, such as the number, location, and characteristics of significant coronary lesions. The score ranges from a minimum of 0 (indicating no significant coronary artery disease) to no fixed maximum (though scores typically do not exceed 100 in clinical practice, with higher values reflecting more extensive disease).
  Scores on a scale | 19.5 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority Comparison of Patient-oriented Composite Endpoint (PoCE) of BiOSS LIM C to a Pre-specified Objective Performance Goal (OPC).
Description: POCE defined as a composite measure of: All-cause mortality, Stroke (Modified Ranking Scale (mRS) ≥1), Any Myocardial infarction (MI) (includes non target vessel territory), Any unplanned revascularization for ischemia (includes all target and nontarget vessels). OPC based on data collected in Excel-study. The safety and efficacy of the BiOSS LIM C® stent with respect to a PoCE at 12 months in a real world LM bifurcation population compared with a pre-specified performance goal was not confirmed. The POLBOS LM study showed that the BiOSS LIM C® stent was not non-inferior to the XIENCE stent for percutaneous treatment of the LM disease.
Time Frame: 12 months
Population: Intention-to-treat population
Measure: Number; unit: Percentage of participants
Groups:
- BiOSS LIM C Arm: Experimental arm
Arm/Group | BiOSS LIM C Arm
Number analyzed (Participants) | 130
Percentage of participants | 38.0

2. Secondary Outcome: Patient-oriented Composite Endpoint (PoCE)
Description: PoCE is defined as a composite of all-cause death, stroke, any MI, and any revascularization
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 38.0

3. Secondary Outcome: Target Vessel Failure
Description: Target Vessel Failure is defined as the composite of cardiac death, target vessel MI, and clinically indicated target vessel revascularization
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 28.5

4. Secondary Outcome: Target Lesion Failure
Description: Target Lesion Failure is defined as a composite of cardiac death, target vessel MI, and clinically indicated target lesion revascularization
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 27.7

5. Secondary Outcome: Mortality
Description: Occurrence of death of any cause
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 1.6

6. Secondary Outcome: Stroke
Description: Occurrence of stroke (with a modified Rankin Scale >=1)
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 1.6

7. Secondary Outcome: Myocardial Infarction
Description: Occurrence of myocardial infarction
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 19.0

8. Secondary Outcome: Revascularization
Description: Occurrence of any revascularization (percutaneous coronary intervention or coronary artery bypass grafting)
Time Frame: 12 months
Population: Intention-to-treat
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 20.3

9. Secondary Outcome: Stent Thrombosis
Description: Occurrence of any stent thrombosis according to standard definitions provided by the Academic Research Consortium
Time Frame: 12 months
Population: Intention-to-treat population
Measure: Number; unit: Percentage of participants
Arm/Group | BiOSS LIM C
Number analyzed (Participants) | 130
Percentage of participants | 0.8

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 months.
Description: Only severe adverse events were captured systematically.
Arm/Group | BiOSS LIM C
All-Cause Mortality (participants affected / at risk) | 2/130
Serious Adverse Events (participants affected / at risk) | 43/130
Other Adverse Events (participants affected / at risk) | 0/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BiOSS LIM C (N=130)
Abnormal liver function (Hepatobiliary disorders) | 1 (1)
Acute pulmonary edema (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Atrial arrhythmia (Cardiac disorders) | 2 (2)
Bleeding (Blood and lymphatic system disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 3 (3)
Coronary stenosis (Cardiac disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 2 (2)
Heart failure (Cardiac disorders) | 2 (2)
In-stent restenosis (Cardiac disorders) | 26 (26)
Low ejection fraction (Cardiac disorders) | 1 (1)
Medication error (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 9 (9)
Pericardial effusion (Cardiac disorders) | 2 (2)
Phlebitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The original sample was intended at 260 but the study only enrolled 130 participants since it was terminated prematurely due to COVID-19, safety concerns, and discontinuation of financial support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03508219/Prot_SAP_000.pdf